CLINICAL TRIAL: NCT00835900
Title: Extended Varenicline for Smoking Cessation: A Pilot Study
Brief Title: An Alternative Dosing Schedule of Varenicline for Smoking Cessation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: I 136208; Pfizer IIR-GA30523; NCT00957515 (obsolete NCT alias)
Record Dates: First submitted 2009-02-03; First posted 2009-02-04 (Estimated); Results first posted 2017-05-30 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-04

CONDITIONS: Smoking Cessation
Keywords: smoking cessation; varenicline; smoking cessation treatment
MeSH Terms: conditions — Smoking Cessation | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- varenicline (Experimental): drug plus counseling.
  Interventions: Drug: varenicline
- placebo (Active Comparator): placebo plus counseling
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: varenicline — variable dosing schedule
  Other Names: Chantix
  Arms: varenicline
Drug: placebo — placebo
  Arms: placebo

SUMMARY:
The purpose of this study is to explore the use of an prolonged alternative dosing schedule using varenicline for smoking cessation leading to greater quit rates and higher rates of continuous abstinence.

DETAILED DESCRIPTION:
This pilot study will utilize a two group randomized design. Adult smokers who are motivated to quit smoking will be randomized to one of two treatment groups. Both groups will receive brief support counseling. During a one-week baseline and the 4-week pre-quit period smoking rate, smoking satisfaction, withdrawal, and craving will be assessed on a daily basis.

ELIGIBILITY:
Inclusion Criteria:

* currently smoking at least 15 cigarettes daily
* in good health
* able to read and speak English fluently
* have a home telephone and plan to reside in Western New York for 6 months
* willing to make quit attempt
* signed informed consent
* who planned quit attempt.

Exclusion Criteria:

* serious medical condition
* depression or mental health condition requiring treatment in the past year
* history of panic disorder, psychosis, bipolar disorder
* alcohol or drug abuse in the past year
* use of tobacco products other than cigarettes
* current use of other cessation pharmacotherapies
* pregnancy/planned pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-03; Primary Completion 2010-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin C Mahoney, MD, PhD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

REFERENCES:
- [Derived] Livingstone-Banks J, Fanshawe TR, Thomas KH, Theodoulou A, Hajizadeh A, Hartman L, Lindson N. Nicotine receptor partial agonists for smoking cessation. Cochrane Database Syst Rev. 2023 May 5;5(5):CD006103. doi: 10.1002/14651858.CD006103.pub8. PMID 37142273

RESULTS

PARTICIPANT FLOW:
Groups:
- Extended Run-In: The Extended run-in group received 4 weeks of varenicline pre-TQD, then continued with standard (11 weeks) post-quit treatment.
- Standard Run-In: The Standard run-in group received 3 weeks of placebo, followed by standard dosing: 1-week pre-TQD varenicline and 11-week post-TQD varenicline, totaling 12 weeks.
  Both groups received brief cognitive-behavioral counseling.
Period: Overall Study
Arm/Group | Extended Run-In | Standard Run-In
Started | 32 | 28
Completed | 27 | 22
Not Completed | 5 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Extended Run-In | Standard Run-In | Total
Number analyzed (Participants) | 32 | 28 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 48 (10) | 49 (10) | 48 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 17 | 35
  Male | 14 | 11 | 25
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Nonwhite | 3 | 5 | 8
  White | 29 | 23 | 52
Baseline CPD [Mean (Standard Deviation); unit: Cigarettes Per Day] | 21 (5) | 21 (5) | 21 (5)

OUTCOME MEASURES:

1. Primary Outcome: Change in Smoking Behavior
Description: Change in cigarettes per day from Week 2 to Week 5
Time Frame: Change in cigarettes per day from Week 2 to Week 5
Population: ITT
Measure: Mean (Standard Error); unit: Change in Cigarettes Per Day
Arm/Group | Extended Run-In | Standard Run-In
Number analyzed (Participants) | 32 | 28
Change in Cigarettes Per Day | -6.3 (0.9) | -3.2 (0.7)

2. Secondary Outcome: Rates of Smoking Cessation.
Description: To parallel most clinical trials of varenicline, we focused on CO-verified (<11 parts per million) continuous abstinence (not even one puff) during the final 4 weeks of treatment (i.e., post-quit weeks 8 through 11). Participants lost to follow-up were coded as smokers.
Time Frame: 12 weeks after quit date.
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Extended Run-In | Standard Run-In
Number analyzed (Participants) | 32 | 28
Participants | 17 | 11

ADVERSE EVENTS:
Arm/Group | Extended Run-In | Standard Run-In
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/32 | 1/28
Other Adverse Events (participants affected / at risk) | 18/32 | 6/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Extended Run-In (N=32) | Standard Run-In (N=28)
Irritability (Psychiatric disorders) | 0 (0) | 1 (1) — One participant in the Standard run-in arm who reported feelings of hostility and irritability 3 weeks after being started on varenicline
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Extended Run-In (N=32) | Standard Run-In (N=28)
Nausea (Gastrointestinal disorders) | 18 (18) | 6 (6)
Constipation (Gastrointestinal disorders) | 8 (8) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No